CLINICAL TRIAL: NCT01269099
Title: Hypokalemia and Intravenous Patient Controlled Analgesia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul Medical Center (Other)
Responsible Party: Won Ho Kim M.D., Seoul Medical Center
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SMC-2010-01-24
Record Dates: First submitted 2010-12-30; First posted 2011-01-04 (Estimated); Last update posted 2011-01-04 (Estimated); Status verified 2010-12

CONDITIONS: General Anesthesia; Laparoscopic Cholecystectomy
Keywords: hypokalemia; intravenous patient controlled analgesia
MeSH Terms: conditions — Hypokalemia | interventions — Analgesia, Patient-Controlled; Fentanyl

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (Active Comparator): Control-group
  Interventions: Drug: Control
- IV-PCA (Experimental): IV-PCA group
  Interventions: Drug: IV-PCA

INTERVENTIONS:
Drug: IV-PCA — IV-PCA (fentanyl 10 mcg/ml) Dose bolus-lock out time - basal = 1.5 ml - 15 min - 1.5 ml/hr
  Other Names: fentanyl
  Arms: IV-PCA
Drug: Control — control group (No-PCA group)
  Other Names: no drug
  Arms: Control

SUMMARY:
The increase in stress hormone level and hyperventilation caused by the postoperative pain may contribute to the development of hypokalemia during postoperative period. Therefore, if the postoperative pain is well controlled by the IV-PCA,the plasma potassium level during the postoperative period may be not affected by stress response. The researchers tried to investigate the effect of IV-PCA on potassium regulation during the postoperative period.

DETAILED DESCRIPTION:
Intravenous patient controlled analgesia(IV-PCA) has been widely used to control postoperative pain. The increase in stress hormone level and hyperventilation caused by the postoperative pain may contribute to the development of hypokalemia during postoperative period. Hypokalemia is a risk factor for postoperative arrhythmia. Therefore, if the postoperative pain is well controlled by the IV-PCA, the plasma potassium level during the postoperative period may be not affected by stress response, and the incidence of hypokalemia may be reduced. The researchers tried to investigate the effect of IV-PCA on potassium regulation during the postoperative period.

The researchers divided the patients undergoing laparoscopic cholecystectomy into two groups of IV-PCA group and control group. The researchers compared the plasma potassium concentration from the preoperative to postoperative period.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing laparoscopic cholecystectomy
* ASA class I or II

Exclusion Criteria:

* Any patients with plasma aldosterone, or glucocorticoid disorder including primary hyperaldosteronism, renovascular hypertension, rennin-secreting tumor, salt-wasting renal disease, Cushing syndrome
* Patients with recent exogenous steroid administration or previous diuretics therapy

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2010-01; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
plasma potassium concentration | one day interval (average)
  blood sample for electrolyte including plasma potassium concentration checking six times
  ; at outpatient department (T1), at 08:00 A.M. of the day of surgery (T2), one hour after the end of surgery (T3), at 8:00 A.M. of first (T4), second (T5), and third postoperative day (T6)

SECONDARY OUTCOMES:
Visual Analogue Scale (VAS) score | one day interval (average)
  patient-reported VAS score during postoperative period checking fourtimes
  ; one hour after the end of surgery (T3), at 8:00 A.M. of first (T4), second (T5), and third postoperative day (T6)

CONTACTS AND LOCATIONS:
Overall Officials: Won Ho Kim, M.D., Principal Investigator — Seoul Medical Center
Locations (1):
- Seoul Medical Center, Seoul, South Korea